CLINICAL TRIAL: NCT03987633
Title: EMPOWER-1: A Multi-site Clinical Cohort Study to Reduce Health Inequality: Identifying Ethnic Disparities in Treatment Failures for Medicines Prescribed to Treat Diseases That Cause Significant Mortality and Morbidity in the UK Population
Brief Title: EMPOWER-1: A Multi-site Clinical Cohort Research Study to Reduce Health Inequality
Acronym: EMPOWER
Status: Recruiting | Type: Observational
Sponsor: Future Genetics Limited (Other)
Responsible Party: Sponsor
Other Study IDs: EMPOWER-1
Record Dates: First submitted 2019-06-12; First posted 2019-06-17 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Atrial Fibrillation; Coronary Heart Disease; Cardiovascular Diseases; Heart Failure; Hypertension; Peripheral Arterial Disease; Stroke, Ischemic; Asthma; Chronic Obstructive Pulmonary Disease; Obesity; Cancer; Chronic Kidney Diseases; Diabetes Mellitus; Dementia; Depression; Epilepsy; Mental Health Disorder; Rheumatoid Arthritis; Blood Pressure; Breast Cancer Risk; Prostate Cancer; Lung Cancers
Keywords: genetic disparity; health inequality; genetics; health outcomes; equality
MeSH Terms: conditions — Atrial Fibrillation; Coronary Disease; Cardiovascular Diseases; Heart Failure; Hypertension; Peripheral Arterial Disease; Ischemic Stroke; Asthma; Pulmonary Disease, Chronic Obstructive; Obesity; Neoplasms; Renal Insufficiency, Chronic; Diabetes Mellitus; Dementia; Depression; Epilepsy; Mental Disorders; Arthritis, Rheumatoid; Prostatic Neoplasms; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva. Where practical, blood or other biological samples may also be voluntarily provided by the patient.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Displaying trait of interest: There are 19 disease areas under investigation. Enrolled patients are segmented into cohorts based on data collected through questionnaires and medical histories. This data-driven approach does not allow for precisely predefined cohorts for the diseases under investigation. Therefore, as a default, the two general predefined cohorts are set as either displaying or not displaying a trait that would form the basis of an investigation.
- Not displaying trait of interest: Please see above.

SUMMARY:
Health inequality and genetic disparity are a significant issue in the United Kingdom (UK).

This study focuses on diseases that are associated with significant morbidity and mortality in the UK, and specifically examines the extent and basis of treatment failure in different patient populations.

The vast majority of drug registration clinical trials have under-representation of ethnic minority populations. In addition, the wider Caucasian populations have reasonably different clinical characteristics to the population that participated in the drug licencing clinical trials. A consequence of this is that drugs are licensed for use in real-world general patient populations where the clinical trial results are simply not statistically significant to specifically demonstrate efficacy or safety in populations that were either absent or under-represented in the drug registration clinical trials. When these facts are considered alongside data that supports significant under-reporting of adverse events in the real-world setting within the UK (and globally, e.g the USA and Europe), it highlights that pharmacovigilance systems are unable to capture drug effectiveness and safety data in a manner that can reasonably assure appropriate prescribing in the wider patient populations.

This large real-world research study aims to identify whether commonly prescribed drugs are effective in treating illnesses that cause significant poor health and death in the different patient populations that represent the UK.

The goal of this study is to generate large quantitative data-sets that may inform clinical practice to reduce the existing health inequality and genetic disparity in the UK.

DETAILED DESCRIPTION:
This multi-centre real-world study will recruit patients across different National Health Service (NHS) sites based in England, where the overall patient population demographic profile is sufficiently variable to allow for meaningful representation of different ethnicities in the analysis of pooled data-sets.

The study addresses the issue of health inequality and genetic disparity in the United Kingdom (UK) by recruiting up to 200,000 patients primarily from the three main ethnic groups in the UK; namely White (Caucasian), African-Caribbean (Black), and South Asian (Asian) populations on a 1:1:1 ratio.

Biological samples, medical records, alongside specific questionnaires will be used in data analyses to help identify treatment failures in different populations for the 19 disease areas under investigation, which are a significant cause of morbidity and mortality in the UK.

Analysis of patient populations may provide real-world evidence around disease prevalence between and within different ethnic groups. The data may also support hypothesis driven genetic analysis to identify putative bio-markers associated with treatment failure.

Data from this study will be published, and findings could better inform clinical practice in the management of diseases that cause significant poor health and death in the different populations that represent the UK.

ELIGIBILITY:
Inclusion Criteria:

1. Patients or their relative/family member is diagnosed with the illness being investigated by this study.
2. All NHS patients that are associated with a participating study site, but do not fall under the first bullet point above, may participate with a view that they may potentially contribute to a case control population in the research study.
3. Subjects agree to:

   1. Gift biological samples, i.e. saliva. Where practical, blood or other biological samples may be voluntarily provided by the patient.
   2. Provide Consent for access to medical records.
   3. Complete disease specific, quality of life, and study associated questionnaires.

Exclusion Criteria:

1. Patient does not provide a valid consent for study participation.
2. Patient is not registered with the NHS for care.
3. Patient lacking capacity, who does not have an illness that is being specifically investigated by this clinical research study.
4. Person lacks capacity and where the personal consultee has not advised that the Person may enrol, in accordance with the Mental Health Act 2005.

Min Age: 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Individuals who are registered as UK NHS patients.
Sampling Method: Non-Probability Sample
Enrollment: 200000 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2028-02-01 (Estimated); Study Completion 2030-02-01 (Estimated)

PRIMARY OUTCOMES:
Ethnic disparities in treatment failure | Ongoing review of data, anticipated completion of primary outcome analysis 4 years post launch
  Identify ethnic disparities in treatment failures for any of the 19 disease states under investigation. The primary outcome is treatment failure, as measured by the discontinuation of a treatment regimen by a clinician in the absence of the cure of the disease, for the most common treatment in each of the 19 diseases.

SECONDARY OUTCOMES:
Ethnic disparities in disease incidence | Ongoing review of data, anticipated completion of analysis 5 years post launch
  Identifying ethnic disparities in disease incidence. The corresponding secondary outcome measure for this is, for each of the 19 diseases under consideration, the diagnosis of the disease. We will use time to diagnosis to examine ethnic disparities in incidence.
Identification of candidate genetic variants associated with observed disparities in treatment failure. | Ongoing review of data, anticipated completion of analysis 5 years post launch
  Another secondary outcome is identifying candidate genetic variants that may underpin observed disparities in treatment failure, for treatments in the 19 diseases under consideration. The corresponding secondary outcome measures used for this are genotypes as identified through whole genome sequencing (WGS) of patient saliva or peripheral blood that are associated with the phenotypes corresponding to the treatment failure previously described as the primary outcome measure.

CONTACTS AND LOCATIONS:
Overall Officials: Dr Mohammed Kamran, Study Director — Future Genetics Limited
Locations (1):
- Future Genetics, The Science Centre, Wolverhampton Science Park, Wolverhampton, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: FUTURE GENETICS website — https://futuregenetics.co.uk/